CLINICAL TRIAL: NCT02165332
Title: A Two-part, Single-center, Single-dose, Randomized, Double-blind, Double-dummy, Placebo-controlled, Positive-controlled, Four-way Crossover Study to Investigate the Effect of RO7033877 on the QT/QTc Interval in Healthy Subjects
Brief Title: A Two-part, Single-dose, Randomized Study to Evaluate the Safety of Supra-therapeutic Doses of RO7033877 and to Investigate the Effect of RO7033877 on the QTc Interval
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: NP29334
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Part 1: Placebo (Placebo Comparator): Saline solution, given as a minimum of a 2 hour infusion
  Interventions: Drug: Part 1: SAD placebo
- Part 1: RO7033877 (Experimental): Single ascending dose
  Interventions: Drug: Part 1: SAD RO7033877
- Part 2: RO7033877 (Experimental): Single-dose 4-way crossover
  Interventions: Drug: Part 2: Treatment A, RO7033877; Drug: Part 2: Treatment B, RO7033877; Drug: Part 2: Treatment C, moxifloxacin; Drug: Part 2: Treatment D, RO7033877 and moxifloxacin placebo

INTERVENTIONS:
Drug: Part 1: SAD RO7033877 — Single dose
  Arms: Part 1: RO7033877
Drug: Part 1: SAD placebo — Single dose
  Arms: Part 1: Placebo
Drug: Part 2: Treatment A, RO7033877 — Single dose RO7033877 and moxifloxacin placebo
  Arms: Part 2: RO7033877
Drug: Part 2: Treatment B, RO7033877 — Single dose RO7033877 and moxifloxacin placebo
  Arms: Part 2: RO7033877
Drug: Part 2: Treatment C, moxifloxacin — Single dose moxifloxacin and RO7033877 placebo
  Arms: Part 2: RO7033877
Drug: Part 2: Treatment D, RO7033877 and moxifloxacin placebo — Single dose moxifloxacin placebo and RO7033877 placebo
  Arms: Part 2: RO7033877

SUMMARY:
This is a two-part study to evaluate the safety and tolerability of supratherapeutic doses of RO7033877 (Part 1) and to investigate the effect of RO7033877 on the QTc interval in healthy volunteers (Part 2). Part 1 is a single ascending dose, randomized, observer-blind, placebo-controlled study to determine the safety tolerability and pharmacokinetics of a supratherapeutic dose to be used in Part 2. Participants will be randomized in up to 8 cohorts to receive a single dose of either RO7033877 or placebo. Part 2 will be a single dose, randomized, double-blind, double dummy, placebo-controlled, positive control, 4-way crossover study. Part 2 will evaluate whether a single therapeutic or supratherapeutic dose of RO7033877 has a threshold pharmacologic effect on cardiac repolarization, as detected by changes in the QT/QTc interval measured by electrocardiogram (ECG). Pharmacokinetic parameters will be assessed for Parts 1 and 2, continuous ECG recordings will be evaluated in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female of non-childbearing potential participants, 18 to 65 years of age, inclusive
* Healthy status is defined as the absence of evidence of any clinically significant, active, or chronic disease following a detailed medical and surgical history, a complete physical examination and vital signs, 12-lead ECG, hematology, blood chemistry, serology and urinalysis and confirmed by a creatinine clearance estimated by formula of Cockcroft-Gault > 80 mL/min/1.73 m2
* Postmenopausal or surgically sterile females (bilateral oophorectomy or hysterectomy performed at least 6 months prior to study participation)
* A body mass index (BMI) between 18 and 30 kg/m2 inclusive and minimum body weight >/= 50 kg, inclusive
* For men with a female partner(s) of childbearing potential: agreement to use a barrier method of contraception during the treatment period and for at least 3 months after the last dose of study drug
* Participants who are non-smokers, or former smokers who have not smoked for at least 45 days prior to screening (former smokers are to have a total of < 10 pack year smoking history)

Exclusion Criteria:

* Women of childbearing potential
* Pregnant or lactating women
* Men with female partners who are lactating or are pregnant
* History of any clinically significant disease, e.g. gastrointestinal, renal, hepatic, cardiovascular, endocrine, hematologic or allergic disease(s), metabolic disorder, cancer (may have had basal or squamous cell carcinoma of skin or cervix as long as surgically removed or deemed cured by cryotherapy, laser therapy, conization, etc., with stability for the past 2 years)
* Any major illness within one month before the first dose of study drug or any febrile illness within one week prior to screening and up to first dose administration
* Any prescribed medications taken within 4 weeks prior to first dosing or within 5 times the elimination half-life of the medication prior to first dosing (whichever is longer)
* Any preparations containing St. John's Wort taken within 4 weeks prior to first dosing
* Any other over-the-counter medications, including vitamins or herbal remedies, taken within 14 days prior to first dosing or within 5 times the elimination half-life of the medication prior to first dosing (whichever is longer); acetaminophen is the only exception
* Taking any nutrients known to modulate cytochrome P450 (CYP) 3A activity. Participants will be instructed to abstain from consuming grapefruit, Seville oranges, and grapefruit- or Seville orange-containing products within 2 weeks prior to administration of study drugs
* Regular consumption of large amounts of caffeine or xanthine-containing substances (e.g. >/= 5 cups of coffee/day, tea, cola, Mountain Dew, chocolate, diet pills, "energy drinks" or any other type of stimulant) or unable to refrain from consumption of caffeine or xanthine-containing substances from 72 hours prior to each entry in the clinic and during the in-house periods
* Any medication that inhibits active tubular secretion (e.g. probenecid, H2 receptor antagonists, trimethoprim) within 4 weeks prior to first dosing
* Participation in an investigational drug or device study within 60 days prior to screening
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* History and/or family history of cardiac anomalies, e.g. congenital long QT syndrome, unexplained syncope, or clinically significant abnormal ECG
* ECG evidence at screening or baseline of, e.g. atrial fibrillation, atrial flutter, complete right or left bundle branch block and/or clinically relevant prolongation of the PR interval as determined by the Investigator

Exclusion criteria for Part 2 only:

* History of allergy or sensitivity to moxifloxacin or other fluoroquinolones, and/or history of tendon rupture when taking or considered time-wise related to consumption of a fluoroquinolone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Part 1: Incidence of adverse events (AEs) after single, supratherapeutic dose of RO7033877 | Up to 30 days
Part 1: Pharmacokinetic parameters derived from plasma and urine concentrations, single dose of RO7033877: Area under the curve (AUC) | Day 1
Part 2: Continuous, 12-lead Holter electrocardiogram (ECG) recordings | Day -1 and 1 of each Period

SECONDARY OUTCOMES:
Incidence of AEs after single IV infusion of RO7033877 | Up to 9 weeks
Part 2 only: Changes in other ECG parameters, descriptive analysis | Up to 9 weeks
Part 2 only: Changes in PK/PD relationships between any effect on ECG and RO7033877 plasma concentrations, descriptive analysis | Up to 9 weeks
Part 2: Area under the concentration-time curve (AUC) of RO7033877 | Day 1 of each Period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Lenexa, Kansas, United States